CLINICAL TRIAL: NCT04589663
Title: An Open-label, Two-period, Single-sequence, Crossover Study to Compare the Systemic Exposure of a Single Inhaled Dose of Mometasone Furoate (MF) When Administered Alone Via the MF Twisthaler® (TH) to a Single Inhaled Dose of QMF149 Indacaterol Acetate/MF Fixed Dose Combination When Administered Via the Concept 1 (C1) Breezhaler® Device in ≥ 6 to < 12 Year Old Asthma Patients
Brief Title: Study to Compare the Pharmacokinetics of Mometasone Furoate Alone and in Combination With Indacaterol in Patients ≥ 6 to < 12 Years Old With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQMF149G2203; 2020-002036-78 (EudraCT Number)
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Asthma
Keywords: QMF149; mometasone furoate; indacaterol; pediatric; asthma; PK
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; QMF149; Standard of Care

STUDY DESIGN:
Intervention Model Description: Single-sequence crossover study
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MF followed by QMF149 (Experimental): Single inhaled dose of mometasone furoate on Day 1 delivered via TH inhaler followed by 4-7 days of washout. On Day 6-9, single inhaled dose of QMF149 delivered via C1 inhaler.
  Interventions: Drug: Mometasone furoate; Drug: QMF149; Drug: Standard of Care (Soc)

INTERVENTIONS:
Drug: Mometasone furoate — Single inhaled dose of 100 µg mometasone furoate (MF) administered via Twisthaler® on Day 1
  Other Names: MF
Drug: QMF149 — Single inhaled dose of QMF149 (75/40 µg indacaterol acetate/MF fixed dose combination) administered via Concept 1 device on Day 6-9
Drug: Standard of Care (Soc) — Asthma therapy: budesonide and salbutamol being the most frequently used (excluding MF and indacaterol acetate)

SUMMARY:
This clinical study was designed to assess the pharmacokinetics, safety and tolerability of single inhaled doses of mometasone furoate (MF) when administered alone via MF Twisthaler® (TH) or as an indacaterol acetate/MF fixed dose combination (QMF149) via the Concept 1 (C1) device in pediatric asthma patients.

DETAILED DESCRIPTION:
This study was an open-label, two-period, single-sequence crossover study that consisted of four distinct study periods:

* Screening: Participants underwent a screening period of up to 14 days where were assessed for eligibility.
* First Treatment: On the first treatment visit (Day 1) participants received a single inhaled dose of 100 μg MF administered via the TH device followed by a 4-7-day washout period.
* Second Treatment: On the second treatment visit (Day 6-9) participants received a single inhaled dose of 75/40 μg indacaterol acetate/MF fixed dose combination (FDC) (QMF149) via C1 (Breezhaler®) device. Participants were allowed to use rescue medication (as needed) and potentially their Standard of Care (SoC) asthma therapy (excluding MF and indacaterol acetate).
* Safety Follow-up: Upon completion of the treatment period, participants were followed up for safety assessments for 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female children ≥ 6 years and < 12 years at the time of study entry.
2. Written informed consent by parent(s)/legal guardian(s) for the pediatric patient and assent by the pediatric patient (depending on local requirements) must be obtained before any study-specific assessment is performed.
3. Confirmed documented diagnosis of asthma, as defined by national or international asthma guidelines for at least 6 months prior to study enrollment.
4. Patients using low dose ICS as asthma controller therapy for at least 4 weeks prior to first treatment.
5. Patients who are familiar with the use of an inhaler device.
6. Patients must be able to comply with the Study Visit Assessment Schedule which includes approximately 7 hours on two occasions, and agree to blood draws as scheduled.
7. Parents/ legal guardian must be willing and able to attend study visits and assist the child with the procedures outlined in the protocol

Exclusion Criteria:

1. Use of other investigational drugs within 5 half-lives of enrollment, or [within 30 days (for small molecules) /until the expected PD effect has returned to baseline (for biologics)], whichever is longer.
2. Patients with weight < 17kg at screening.
3. Patients currently taking MF products for any reason at least 7 days prior to Day 1. Patients can enroll if MF was discontinued at least 7 days prior to Day 1 and MF is substituted with a different steroid during entire study duration to avoid its potential impact on PK assessment. These MF products include inhalation, topical and/or nasal spray formulations.
4. Patients on medium- and high- dose ICS or any dose ICS/LABA combination.
5. Patients taking maintenance controller therapy (eg LABAs and theophylline) within 4 weeks of screening or during the study. LTRAs are permitted provided that patients have been on a stable dose for 4 weeks prior to screening. Patients using short-acting bronchodilators on occasional basis as rescue medication can enroll, however, these medications must be withheld at least 8 hours prior to study dosing visits and during PK sampling.
6. Contraindicated for treatment with, or having a history of reactions/hypersensitivity to any of the following inhaled drugs, drugs of a similar class, or any component there of:

   * Adrenoreceptor agonist agent Lactose or any of the other excipients of the study drug (including patients with history of galactose intolerance, lactase deficiency or glucose-galactose malabsorption)
   * Corticosteroids
   * Indacaterol and/or MF
7. History of chronic lung disease other than asthma within 3 months of first treatment visit (Day 1), cystic fibrosis, mycobacterial or other infection (including active SARS-CoV-2, tuberculosis or atypical mycobacterial disease).
8. History of active bacterial, viral or fungal infection (including SARS-CoV-2) within 6 weeks of first treatment visit (Day 1).
9. Patients who have had an asthma attack/exacerbation requiring systemic steroids or hospitalization or emergency room visit within 6 weeks of first treatment visit (Day 1).
10. Patients who, in the opinion of the investigator, are not able to comply with study treatment or who have any medical or mental disorder, situation, or diagnosis, which could interfere with the proper completion of the study protocol requirements or pose a safety risk while participating in the study.
11. Parent/guardian has a history of psychiatric disease, intellectual deficiency, substance abuse, or other condition (e.g. inability to read, comprehend and write) which will limit the validity of consent for their child to participate in this study.
12. Hemoglobin levels outside normal ranges at screening.
13. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the patient in case of participation in the study.
14. Patients who have a clinically significant ECG abnormality or clinically significant abnormal lab values reported at Screening Visit.
15. Patients with a history of long QT syndrome or whose corrected QT interval (QTc) measured at Screening Visit (Fridericia method) is prolonged (≥ 450 msec for males and females 6 - 12 years old).
16. Use of any prescription drugs, herbal supplements, prescribed medicinal use of cannabis/marijuana, within four weeks prior to initial dosing, and/or over-the-counter (OTC) medication, dietary supplements within two weeks prior to initial dosing. If needed, (i.e. an incidental and limited need) paracetamol/acetaminophen is acceptable, but must be documented in the Concomitant medications / Significant non-drug therapies page of the CRF.
17. History of malignancy of any organ system, treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
18. Patient is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
19. Pregnant or nursing (lactating) females.
20. Inability to properly train in the use of the In-Check DIAL® at screening (at the investigator's discretion).
21. Inability to properly train in the use of the Twisthaler® or Concept 1 Breezhaler® prior to dosing (at the investigator's discretion).
22. History of paradoxical bronchospasm in response to inhaled medicines.
23. Patients receiving any medications in the classes specified in protocol Table 6-2 unless they undergo the required washout period prior to Day 1.
24. Patients who are sexually active.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Novartis Investigative Site, Nagykanizsa, Hungary
- South Africa (2):
  - Novartis Investigative Site, George, Western Cape
  - Novartis Investigative Site, Cape Town

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 sites in 2 countries
Pre-assignment Details: Participants underwent a Screening period of up to 14 days
Period: Overall Study
Arm/Group | MF Followed by QMF149
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MF Followed by QMF149
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.0 (1.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 15
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Mometasone Furoate Plasma Concentration (Cmax)
Description: Mometasone furoate plasma concentrations were determined by a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method. Cmax of mometasone furoate was determined with Phoenix WinNonlin (Version 8.0 or higher).
  A correction factor was applied to MF pharmacokinetic parameters to consider the first-dose effect that is based on the fact that the participants in this study received a single dose from single unused (unprimed) C1 and TH devices. Unprimed devices are not coated with the formulation, and therefore may lead to lower fine particle mass (FPM) and delivered dose compared to later doses actuated from the device throughout its use time. The first-dose correction factor (FPMprimed (MF) / FPMunprimed (MF)) for MF delivered via TH was 1.26 and for MF delivered via C1 it was 1.62.
Time Frame: pre-dose, 0.5, 1, 2, 3 and 6 hours post-dose on Day 1 and Day 6-9
Population: The overall number of participants analyzed includes all participants with evaluable data for the endpoint.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- MF 100 ug Via Twisthaler: Single inhaled dose of mometasone furoate on Day 1 delivered via TH inhaler followed by 4-7 days of washout
- QMF149 75/40 ug Via Concept 1: Single inhaled dose of QMF149 delivered via C1 inhaler on Day 6-9
Arm/Group | MF 100 ug Via Twisthaler | QMF149 75/40 ug Via Concept 1
Number analyzed (Participants) | 23 | 24
pg/mL | 51.9 (23.5) | 53.5 (16)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time Point 6h (AUC0-6h) of Mometasone Furoate
Description: AUC0-6h of mometasone furoate was determined using non-compartment methods with Phoenix WinNonlin (Version 8.0 or higher). The linear trapezoidal rule was used for AUC0-6h calculation.
  A correction factor was applied to MF pharmacokinetic parameters to consider the first-dose effect that is based on the fact that the participants in this study received a single dose from single unused (unprimed) C1 and TH devices. Unprimed devices are not coated with the formulation, and therefore may lead to lower fine particle mass (FPM) and delivered dose compared to later doses actuated from the device throughout its use time. The first-dose correction factor (FPMprimed (MF) / FPMunprimed (MF)) for MF delivered via TH was 1.26 and for MF delivered via C1 it was 1.62.
Time Frame: pre-dose, 0.5, 1, 2, 3 and 6 hours post-dose on Day 1 and Day 6-9
Population: The overall number of participants analyzed includes all participants with evaluable data for the endpoint.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | MF 100 ug Via Twisthaler | QMF149 75/40 ug Via Concept 1
Number analyzed (Participants) | 18 | 23
h*pg/mL | 208 (102) | 176 (57.5)

3. Secondary Outcome: Systemic Exposure to Indacaterol in Plasma
Description: Systemic exposure to indacaterol in plasma following sparse pharmacokinetic (PK) sampling on Day 6-9 after inhalation of QMF149.
  A correction factor was applied to indacaterol plasma concentrations to consider the first-dose effect that is based on the fact that the participants in this study received a single dose from single unused (unprimed) C1 and TH devices. Unprimed devices are not coated with the formulation, and therefore may lead to lower fine particle mass (FPM) and delivered dose compared to later doses actuated from the device throughout its use time. The first-dose correction factor (FPMprimed (indacaterol) / FPMunprimed (indacaterol)) for indacaterol delivered via C1 was 2.0.
Time Frame: pre-dose, 0.25 and 1 hour post-dose on Day 6-9
Population: The overall number of participants analyzed includes all participants. The number analyzed per row represents participants with evaluable data at each time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MF Followed by QMF149
Number analyzed (Participants) | 24
pg/mL
  Pre-dose | 0 (0)
  0.25 hours post-dose | 102.0 (54.9)
  1 hours post-dose: number analyzed (Participants) | 22
  1 hours post-dose | 62.3 (26.2)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the start of treatment to 30 days after end of treatment, assessed up to maximum duration of 39 days.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Groups:
- Total: Total
Arm/Group | MF 100 ug Via Twisthaler | QMF149 75/40 ug Via Concept 1 | Total
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 3/24 | 0/24 | 3/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MF 100 ug Via Twisthaler (N=24) | QMF149 75/40 ug Via Concept 1 (N=24) | Total (N=24)
Device failure (Product Issues) | 2 | 0 | 2
Influenza (Infections and infestations) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT04589663/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT04589663/SAP_001.pdf